CLINICAL TRIAL: NCT01790347
Title: The Role of a Supervised Physical Exercise Program as a Alternative on the Control of Maternal Gestational Weight Gain
Brief Title: Physical Exercise Controls Gestational Weight Gain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Madrid (Other)
Responsible Party: Principal Investigator, María Perales Santaella, PhD student, Technical University of Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Gestational weight gain
Record Dates: First submitted 2013-02-04; First posted 2013-02-13 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-01

CONDITIONS: Pregnancy
Keywords: Exercise; Aerobic; Resistance training; Pregnancy; Maternal weight gain; IOM recommendations
MeSH Terms: conditions — Motor Activity; Gestational Weight Gain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise group (Experimental)
  Interventions: Behavioral: Exercise group
- Control group (No Intervention): Sedentary pregnant women

INTERVENTIONS:
Behavioral: Exercise group — The physical conditioning program included a total of three 50-55 minute sessions per week. Pregnant women started at 9 weeks and finished at 38-39 weeks, therefore, an average of 85 training sessions were planned for each participant. All subjects wore a heart rate (HR) monitor (Polar FT7, Finland) during the training sessions to ensure that the exercise intensity was light to moderate.
  Each session included 10 min of warm up and 10 min of cool down which included an specific pelvic floor muscles training. The core section of the exercise session lasted from 25 to 30 min and included moderate-intensity aerobic exercises once a week and resistance exercises twice a week.
  Arms: Exercise group

SUMMARY:
An estimated two-thirds to three- quarters of women experience gestational weight gain outside of IOM's 2009 recommendations: 40-60% of women experiencing excessive gain and 15-30% inadequate gain. Not gaining the adequate weight gain is strongly associated with several maternal and fetal complications..

DETAILED DESCRIPTION:
The aim of this study was to assess the role of a supervised exercise programme on the control of maternal gestational weight gain and its consequences.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy and able to exercise following American College of Obstetricians and Gynecologists (ACOG) guidelines
* Being able to communicate in spanish

Exclusion Criteria:

* Obstetrician complications
* Being interested in the study after 18 weeks
* Not being regular in physical exercise program
* Younger than 18 years old

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2350 (Actual)
Dates: Start 2007-09; Primary Completion 2011-01 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Maternal gestational weight gain | 40-42 weeks
  Maternal weight gain

SECONDARY OUTCOMES:
Maternal gestational diabetes | From 24 to 26 week
  Gestational diabetes
Fetal body mass index | 38-42 weeks
  Baby body Mass index (BMI)

OTHER OUTCOMES:
Gestational age | 36-42 weeks
  Number of weeks of gestation at labor
Fetal outcome | 36-42 weeks
  Type of labor

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Barakat, PhD, Study Director — Universidad Politecnica de Madrid
Locations (1):
- Universidad Politécnica de Madrid, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Ruiz JR, Perales M, Pelaez M, Lopez C, Lucia A, Barakat R. Supervised exercise-based intervention to prevent excessive gestational weight gain: a randomized controlled trial. Mayo Clin Proc. 2013 Dec;88(12):1388-97. doi: 10.1016/j.mayocp.2013.07.020. PMID 24290112